CLINICAL TRIAL: NCT03383211
Title: Transcriptomic Profile of the Immune Response to BCG Vaccination in Neonates Born to HIV and LTBI Infected and Non-infected Mothers
Brief Title: Immune Response to BCG Vaccination in Neonates Born to HIV and LTBI Infected and Non-infected Mothers
Acronym: IMMUNEO
Status: Completed | Type: Observational
Sponsor: George Washington University (Other)
Collaborators: Universitatea de Stat de Medicina si Farmacie Nicolae Testemiţanu (Other); Children's National Research Institute (Other); DC-Center for Aids Research (DC-CFAR) (Unknown); SeqLL, Inc. (Unknown)
Responsible Party: Principal Investigator, Ian Toma, MD, PhD, Associate Research Professor, George Washington University
Other Study IDs: GWMDA2017
Record Dates: First submitted 2017-12-19; First posted 2017-12-26 (Actual); Last update posted 2021-10-20 (Actual); Status verified 2021-10

CONDITIONS: HIV Infections; Neonatal Infection; LTBI - Latent Tuberculosis Infection; Immune Tolerance
Keywords: RNAseq; Next Generation Sequencing; Transcriptome; Peripheral blood transcripts; Tempus Blood RNA Tubes
MeSH Terms: conditions — HIV Infections; Latent Tuberculosis | interventions — Base Sequence

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — RNA isolated from peripheral blood.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- HIV+: Pregnant women diagnosed with HIV infection during pregnancy. No intervention beyond the standard care provided for such cohort.
  Interventions: Other: RNAseq
- LTBI: Pregnant women diagnosed with Latent form of TB infection (LTBI). No intervention beyond the standard of care provided for such cohort.
  Interventions: Other: RNAseq
- HV+/LTBI: Pregnant women diagnosed with HIV and LTBI co-infection. No intervention beyond the standard of care provided for such cohort.
  Interventions: Other: RNAseq
- Healthy Control: Healthy pregnant women without HIV or LTBI. No intervention beyond the standard of care provided for such cohort.
  Interventions: Other: RNAseq

INTERVENTIONS:
Other: RNAseq — Transcriptome profiling of peripheral blood using RNA sequencing technology

SUMMARY:
Maternal infections affect the basal immune status of neonates. One of the possible mechanism is the fetomaternal microchimerism, in which some cells and active substances are exchanged bi-directionally between maternal and fetal circulation through placenta. Even in the absence of a direct (vertical) transmission of pathogens to fetuses, certain infections make the neonates more prone to allergies and some adverse events of early vaccinations. We postulate that the basal immune status of neonates born to HIV and LTBI infected mothers is primed by gestational exposure to immunological active molecules, which could results in an altered response to early BCG vaccination. Transcripts expression identified by RNA sequencing are compared between sets of mother-child and their respective umbilical cord blood, and between groups of infected and non-infected pairs.

DETAILED DESCRIPTION:
The study is comparing the transcriptomic profiles of maternal peripheral blood with those of the corresponding umbilical cord blood and neonatal peripheral blood pre- and post-BCG vaccination.

For RNA sequencing, the samples are collected in Tempus RNA Blood tubes at 5 time-points (TP): maternal peripheral blood at the time of initial diagnosis with HIV (first OBGYN consultation @ 12-16 weeks of pregnancy - TP1); repeated HIV test in 3rd trimester of pregnancy (34-36 weeks- TP2); umbilical cord blood (after delivery and ligation- TP3); neonates (24 hours after birth and after HBV vaccination, prior to BCG vaccination- TP4); and neonates (7 days after BCG vaccination- TP5).

As an indicator of the inflammatory status, the peripheral blood samples collected at the same TP are stained for serological markers of inflammation, exhaustion, maturation and activation.

An advanced bioinformatics analysis examines the immune-associated transcripts in RNAseq samples to assess the V(D)J recombination of T-cell and B-cell receptors along with immune-associated SNPs.

The main goal of the study is to identify in umbilical cord blood the genomic biomarkers of the neonatal basal immune status for guiding an optimal BCG immunization protocol for such neonates and to avoid potential adverse events after vaccination.

ELIGIBILITY:
Inclusion Criteria:

Pregnant women, 18-45 years old, capable of reading and understanding the informed consent and the purpose of the study The newborns of the enrolled pregnant women. Women of reproductive age with or without HIV and LTBI infections

Exclusion Criteria:

Pregnant women younger than 18 years or older than 45 years of age Pregnant women and infants with known genetic abnormalities, including primary immunodeficiencies; or receiving immunosuppressive therapy; Infants infected in utero, perinatally, or neonatally with hepatitis B virus, Treponema pallidum (syphilis), Toxoplasma gondii, rubella virus, cytomegalovirus, or herpes simplex virus.

Pregnant women with known history of alcohol or drug abuse, cancer diagnosis and treatment with chemotherapeutic agents, radiation.

Pregnant women with history of organ transplantation.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Pregnant women or women of the reproductive age
Study Population: Pregnant women, 18-45 years old who consented for participation in the study. All women are managed by the local national healthcare system without any interventions from the research team. The collection of samples is performed by the local trained medical personnel, and the samples are processed in a research laboratory.
Sampling Method: Non-Probability Sample
Enrollment: 125 (Actual)
Dates: Start 2017-06-16 (Actual); Primary Completion 2020-09-01 (Actual); Study Completion 2021-06-30 (Actual)

PRIMARY OUTCOMES:
Changes in immune-associated transcripts | Collection of samples 7-days after BCG vaccination
  Identification of transcripts that are differential expressed between groups

CONTACTS AND LOCATIONS:
Overall Officials: Ian Toma, MD, PhD, Principal Investigator — George Washington University
Locations (2):
- Moldova (2):
  - Clinical Municipal Hospital No. 1, Chisinau
  - National Center for Mother and Child Health, Chisinau

IPD SHARING:
Plan to Share IPD: Yes
Genomic data will be submitted to the NCBI SRA archive
Time Frame: Upon completion of analysis
Access Criteria: NCBI standard access criteria